CLINICAL TRIAL: NCT01580696
Title: Phase I/IIa Trial of Folate Binding Protein (FBP) Peptide (E39) Vaccine in Ovarian and Endometrial Cancer Patients
Brief Title: Phase I/IIa Trial of Folate Binding Protein Vaccine in Ovarian Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: COL George Peoples, MD, FACS (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, COL George Peoples, MD, FACS, Chief, Surgical Oncology, Brooke Army Medical Center, Director and Principal Investigator, Cancer Vaccine Development Program, San Antonio Military Medical Center
Organization: San Antonio Military Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 05-20025/20288
Record Dates: First submitted 2012-04-16; First posted 2012-04-19 (Estimated); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Ovarian Cancer; Endometrial Cancer; Fallopian Cancer; Peritoneal Cancer
Keywords: Folate binding protein; E39 vaccine; Stage I-IV ovarian cancer; Stage I-IV endometrial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation study of E39 + GM-CSF in HLA-A2+ patients with HLA-A2- patients followed as a control arm
Oversight: Data Monitoring Committee: No

ARMS (7):
- Non-vaccine clinically matched control group (Active Comparator): HLA-A2-negative patients and HLA-A2+ patients who decline the vaccine will be followed clinically as matched controls for disease recurrence/progression.
  Interventions: Other: Non-vaccine clinically matched control group
- E39 peptide (100mcg)/GM-CSF vaccine plus E39 booster (Experimental): HLA-A2+ patients receive 100mg E39 peptide/GM-CSF vaccine intradermally every 3-4 weeks for a total of up to six inoculations followed by 500mg booster inoculations of E39 6 and 12 months after completion of the primary vaccine series.
  Interventions: Biological: E39 peptide (100mcg)/GM-CSF vaccine plus E39 booster
- E39 peptide (500mcg) /GM-CSF vaccine plus E39 booster (Experimental): HLA-A2+ patients receive 500mg E39 peptide/GM-CSF vaccine intradermally every 3-4 weeks for a total of up to six inoculations followed by 500mg booster inoculations of E39 6 and 12 months after completion of the primary vaccine series.
  Interventions: Biological: E39 peptide (500mcg)/GM-CSF vaccine plus E39 booster
- E39 peptide (1000mcg) /GM-CSF vaccine plus E39 booster (Experimental): HLA-A2+ patients receive 1000mg E39 peptide/GM-CSF vaccine intradermally every 3-4 weeks for a total of up to six inoculations followed by 500mg booster inoculations of E39 6 and 12 months after completion of the primary vaccine series.
  Interventions: Biological: E39 peptide (1000mcg)/GM-CSF vaccine plus E39 booster
- E39 peptide (100mcg)/GM-CSF vaccine plus J65 booster (Experimental): HLA-A2+ patients receive 100mg E39 peptide/GM-CSF vaccine intradermally every 3-4 weeks for a total of up to six inoculations followed by 500mg booster inoculations of E39' (J65) 6 and 12 months after completion of the primary vaccine series.
  Interventions: Biological: E39 peptide (100mcg)/GM-CSF vaccine plus J65 booster
- E39 peptide (500mcg) /GM-CSF vaccine plus J65 booster (Experimental): HLA-A2+ patients receive 500mg E39 peptide/GM-CSF vaccine intradermally every 3-4 weeks for a total of up to six inoculations followed by 500mg booster inoculations of E39' (J65) 6 and 12 months after completion of the primary vaccine series.
  Interventions: Biological: E39 peptide (500mcg)/GM-CSF vaccine plus J65 booster
- E39 peptide (1000mcg) /GM-CSF vaccine plus J65 booster (Experimental): HLA-A2+ patients receive 1000mg E39 peptide/GM-CSF vaccine intradermally every 3-4 weeks for a total of up to six inoculations followed by 500mg booster inoculations of E39' (J65) 6 and 12 months after completion of the primary vaccine series.
  Interventions: Biological: E39 peptide (1000mcg)/GM-CSF vaccine plus J65 booster

INTERVENTIONS:
Biological: E39 peptide (100mcg)/GM-CSF vaccine plus E39 booster — 100mcg lyophilized E39 peptide is suspended in bacteriostatic water for injection in individual cryovials and frozen. At the time of vaccine administration, the suspended peptide is thawed and mixed thoroughly with 250mcg GM-CSF in the syringe. This constitutes the E39 vaccine at this dose.
  Subsequently, patients will receive a booster of E39 dosed at 500mcg and mixed with 250mcg of GM-CSF. The boosters will be given at 6 and 12 months after completing the primary vaccine series above.
  Other Names: E39 peptide (FBP, 191-199, EIWTHSTKV); GM-CSF (sargramostim)
  Arms: E39 peptide (100mcg)/GM-CSF vaccine plus E39 booster
Other: Non-vaccine clinically matched control group — HLA-A2-negative patients or HLA-A2-positive patients who decline the vaccine will be followed clinically as matched controls for disease recurrence/progression. No experimental treatment will be administered to this group.
  Other Names: Clinical tracking for disease progression/recurrence
  Arms: Non-vaccine clinically matched control group
Biological: E39 peptide (500mcg)/GM-CSF vaccine plus E39 booster — 500mcg lyophilized E39 peptide is suspended in bacteriostatic water for injection in individual cryovials and frozen. At the time of vaccine administration, the suspended peptide is thawed and mixed thoroughly with 250mcg GM-CSF in the syringe. This constitutes the E39 vaccine at this dose.
  Subsequently, patients will receive a booster of E39 dosed at 500mcg and mixed with 250mcg of GM-CSF. The boosters will be given at 6 and 12 months after completing the primary vaccine series above.
  Other Names: E39 peptide (FBP, 191-199, EIWTHSTKV); GM-CSF (sargramostim)
  Arms: E39 peptide (500mcg) /GM-CSF vaccine plus E39 booster
Biological: E39 peptide (1000mcg)/GM-CSF vaccine plus E39 booster — 1000mcg lyophilized E39 peptide is suspended in bacteriostatic water for injection in individual cryovials and frozen. At the time of vaccine administration, the suspended peptide is thawed and mixed thoroughly with 250mcg GM-CSF in the syringe. This constitutes the E39 vaccine at this dose.
  Subsequently, patients will receive a booster of E39 dosed at 500mcg and mixed with 250mcg of GM-CSF. The boosters will be given at 6 and 12 months after completing the primary vaccine series above.
  Other Names: E39 peptide (FBP, 191-199, EIWTHSTKV); GM-CSF (sargramostim)
  Arms: E39 peptide (1000mcg) /GM-CSF vaccine plus E39 booster
Biological: E39 peptide (100mcg)/GM-CSF vaccine plus J65 booster — 100mcg lyophilized E39 peptide is suspended in bacteriostatic water for injection in individual cryovials and frozen. At the time of vaccine administration, the suspended peptide is thawed and mixed thoroughly with 250mcg GM-CSF in the syringe. This constitutes the E39 vaccine at this dose.
  Subsequently, patients will receive a booster of J65 dosed at 500mcg and mixed with 250mcg of GM-CSF. The boosters will be given at 6 and 12 months after completing the primary vaccine series above.
  Other Names: E39 peptide (FBP, 191-199, EIWTHSTKV); GM-CSF (sargramostim); J65 peptide (an attenuated peptide of E39, EIWTFSTKV)
  Arms: E39 peptide (100mcg)/GM-CSF vaccine plus J65 booster
Biological: E39 peptide (500mcg)/GM-CSF vaccine plus J65 booster — 500mcg lyophilized E39 peptide is suspended in bacteriostatic water for injection in individual cryovials and frozen. At the time of vaccine administration, the suspended peptide is thawed and mixed thoroughly with 250mcg GM-CSF in the syringe. This constitutes the E39 vaccine at this dose.
  Subsequently, patients will receive a booster of J65 dosed at 500mcg and mixed with 250mcg of GM-CSF. The boosters will be given at 6 and 12 months after completing the primary vaccine series above.
  Other Names: E39 peptide (FBP, 191-199, EIWTHSTKV); GM-CSF (sargramostim); J65 peptide (an attenuated peptide of E39, EIWTFSTKV)
  Arms: E39 peptide (500mcg) /GM-CSF vaccine plus J65 booster
Biological: E39 peptide (1000mcg)/GM-CSF vaccine plus J65 booster — 1000mcg lyophilized E39 peptide is suspended in bacteriostatic water for injection in individual cryovials and frozen. At the time of vaccine administration, the suspended peptide is thawed and mixed thoroughly with 250mcg GM-CSF in the syringe. This constitutes the E39 vaccine at this dose.
  Subsequently, patients will receive a booster of J65 dosed at 500mcg and mixed with 250mcg of GM-CSF. The boosters will be given at 6 and 12 months after completing the primary vaccine series above.
  Other Names: E39 peptide (FBP, 191-199, EIWTHSTKV); GM-CSF (sargramostim); J65 peptide (an attenuated peptide of E39, EIWTFSTKV)
  Arms: E39 peptide (1000mcg) /GM-CSF vaccine plus J65 booster

SUMMARY:
Folate binding protein (FBP) is highly over-expressed in breast, ovarian and endometrial cancers and is the source of immunogenic peptides (E39) that can stimulate cytotoxic T lymphocytes (CTL) to recognize and destroy FBP-expressing cancer cells in the laboratory. The purpose of this study is to test whether a peptide-based vaccine consisting of the E39 peptide mixed with the FDA-approved immunoadjuvant granulocyte macrophage colony-stimulating factor (GM-CSF) is safe and effective at inducing an in vivo peptide-specific immune response. Furthermore, the investigators intend to determine the best dose of the vaccine to utilize to produce this immunity most efficiently. The investigators will determine whether immunity to FBP will prevent clinical recurrence. Additionally, the investigators will compare these results with results from a trial utilizing the E75 peptide (from the HER2/neu protein) in ovarian and endometrial cancer patients in preparation for studying a combination vaccine.

DETAILED DESCRIPTION:
In this study, investigators intend to assess the safety and document local and systemic toxicity to the folate binding protein (FBP) peptide vaccine E39 + GM-CSF given in the adjuvant setting. Investigators also intend to determine the maximum tolerated dose (MTD) and optimal biologic dose (OBD) for the peptide vaccine, as well as evaluate the in vivo cellular immune response to the vaccine. Time to recurrence in the vaccinated patients vs. matched controls will be tracked.

The primary endpoints are the safety and optimal dosing of the vaccine to induce an in vivo peptide-specific immune response. The clinical endpoint is time to recurrence from date of enrollment.

The study will be a multicenter, phase I/IIa trial of the FBP peptide E39 + GM-CSF. The target study population is female civilian and military health care beneficiaries over the age of 18 years with a diagnosis of ovarian, endometrial, fallopian, or peritoneal cancer who have undergone primary surgical and medical therapies, are post-menopausal or have surgically induced menopause, and are currently without evidence of disease. Disease-free subjects after standard of care multi-modality therapy will be screened and HLA typed since the E39 vaccine is specific for HLA-A2+ patients (approximately 40% of the US population). HLA-A2-patients will be followed as prospective clinically matched controls for recurrence.

HLA-A2+ patients who meet all other eligibility criteria will be tested for biomarkers that indicate progression/recurrence of ovarian and advanced uterine cancer FBP. FBP+ and HLA-A2+ patients will be vaccinated with the FBP peptide (E39) and GM-CSF. HLA-A2-negative patients and those individuals who are eligible to receive the vaccine but who decline will be followed clinically as matched controls for disease recurrence/progression.

Treatment will begin within one month of the subject enrollment in the study and confirmation of eligibility. The 1 ml by volume vaccine will be administered intradermally in 0.5 mL inoculums at two different sites within 5 cm of each other. A total of six vaccinations will be given every 3-4 weeks and will be administered in the same lymph node draining area. The dose escalation scheme is for three patients to receive each of the doses: 100, 500, and 1,000 mcg of peptide. Patients will be enrolled consecutively. An additional three patients may receive a given a dose depending on the presence of dose limiting toxicity (DLT). Prior to the fourth vaccination, each patient will be assessed for liver, renal, and hematopoietic function. If organ function is stable and no DLT is seen, then the patient will continue with the series. After the last patient in a given dose group has completed the third inoculation and organ function is proven stable, then the next dose group will be initiated. Optimal biologic dose (OBD) is defined as the minimum dose of the vaccine that gives the most optimal and lasting in vivo immunologic response to the vaccinated peptide. Up to 15 patients will be vaccinated at the OBD.

Additionally, the E39-vaccinated patients will be randomized to receive either E39 or J65 (an attenuated version of E39) as a booster to promote long-term E39-specific immunity. The clinical endpoints are long-term FBP immunity, time to recurrence from date of enrollment and 5-year survival rate. Those individuals who are eligible to receive the vaccine, but who decline and all HLA-A2- patients will be followed clinically as matched controls for disease recurrence/progression

Subjects will be followed for safety issues, immunologic response and clinical recurrence. Subjects will be monitored 48-72 hours after each inoculation for reaction to the inoculation as well as documentation of any adverse effects experienced. Immunologic response will be documented with both ex vivo phenotypic and functional assays as well as in vivo delayed type hypersensitivity (DTH) reactions. All patients will be followed for a total of 5 years to document disease-free status.

The investigators intend to enroll up to 60 patients will be enrolled study-wide (15-24 in the vaccine arm, up to 36 in the control arm). With accrual beginning in April 2012 enrollment of the last patient is anticipated to occur in December 2014 followed by a five-year follow-up period. The duration of the trial is expected to be seven years.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in the study based on the following criteria. (Enrollment may commence 1 month from completion of standard primary therapies and up to two years after completion of treatment.)

1. Ovarian or endometrial, fallopian and peritoneal cancer
2. Completion of primary first-line therapies (i.e., surgery, chemotherapy, immunotherapy and radiation therapy as appropriate per standard of care for patient's specific cancer)
3. Stage I-IV but no evidence of disease (NED) after completion of primary therapies
4. Post-menopausal or rendered surgically infertile
5. HLA-A2+ patients will receive the vaccine; HLA-A2- patients will be eligible to participate in the control group
6. Good performance status (Karnofsky > 60%, ECOG ≤ 2)
7. CBC, CMP, and CA-125 within 2 months of enrollment
8. Capable of informed consent

Exclusion Criteria:

Patients will be excluded from the study based on the following criteria:

1. Receiving immunosuppressive therapy to include chemotherapy, steroids, or methotrexate
2. Not post-menopausal or not rendered surgically infertile
3. Pregnancy
4. In poor health (Karnofsky < 60%, ECOG > 2)
5. Tbili > 1.5, creatinine > 2, hemoglobin < 10, platelets < 50,000, WBC < 2,000
6. Active interstitial lung disease; asthma requiring more than as needed bronchodilators for management; or other autoimmune lung disease
7. Involved in other experimental protocols (except with permission of the other study PI and completion of the other study dosing regimen)
8. History of autoimmune disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-04; Primary Completion 2016-07-31 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
Safety and Local/Systemic Toxicity | Duration of the vaccine series
  Standard local and systemic toxicities will be collected and graded per the National Cancer Institute Common Terminology Criteria for Adverse Events, v4.03 toxicity scale. For the vaccine series (one vaccine/month for six months), patients will be monitored closely for one hour after vaccine inoculation with questioning, serial exams and vital signs every 15 minutes to observe for a hypersensitivity reaction. Patients will also return to the clinic 48-72 hours after each inoculation for questioning regarding systemic toxicity and to examine and measure inoculation site local reactions.

SECONDARY OUTCOMES:
Disease-free survival | Disease-free survival up to 36 months
  Disease-free survival (DFS) for all patients regardless of randomization will be determined by the patients' own physicians at the individual study sites during routine follow-up screening. This will occur every three months for the first 24 months after diagnosis and then every six months for an additional 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: John C Elkas, MD, JD, Principal Investigator — Mid-Atlantic Gynecologic Oncology & Pelvic Surgical Associates; COL George E. Peoples, MD, Study Director — Brooke Army Medical Center
Locations (1):
- Mid-Atlantic Gynecologic Oncology & Pelvic Surgery Associates, Annandale, Virginia, United States